CLINICAL TRIAL: NCT07046351
Title: weSIPsmarter: An Adaptation and Efficacy Trial to Evaluate a Behaviorally Based Digital Health Intervention Aimed at Reducing Sugary Drinks Among Rural Head Start Preschoolers and Their Parents
Brief Title: weSIPsmarter: Evaluating a Digital Health Intervention Aimed at Reducing Sugary Drinks Among Rural Head Start Preschoolers and Their Parents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jamie Zoellner, PhD RD, Professor, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-SBS-6590; R01CA282436 (NIH)
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-11

CONDITIONS: Sugary Beverages

STUDY DESIGN:
Intervention Model Description: Cluster randomized design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- weSIPsmarter (Experimental): weSIPsmarter, targets parents as the agent of change and will be a highly interactive, structured program. It will consist of multiple evidence-based behavioral change components, including use of ecological momentary assessment (EMA) to encourage self-monitoring of beverage behaviors and parenting feeding practices, goal setting and action planning, a resource help line, and drinking water vouchers for families with concerns related to in-home tap water quality. weSIPsmarter participants will be engaged in completing six Cores, tracking daily sugary drink intake for parents and child, and completing daily weigh-ins for parents only.
  Interventions: Behavioral: weSIPsmarter
- weLearn2Read (Other): weLearn2Read participants will be engaged in completing six Cores. Participants will also receive 6 children's books, matched to each Core, which will be mailed to the participants' homes. Parents in the weLearn2Read control can also opt to receive reminders (email or text) to encourage reading readiness.
  Interventions: Behavioral: weLearn2Read

INTERVENTIONS:
Behavioral: weSIPsmarter — weSIPsmarter is grounded by the Theory of Planned Behavior as well as Satter's Feeding Dynamic Model. weSIPsmarter will also integrate relevant behavior change techniques and target concepts from health literacy, health numerary, media literacy, and eHealth literacy.
  Arms: weSIPsmarter
Behavioral: weLearn2Read — weLearn2Read participants will have access to a website with resources to improve reading readiness, including 6 structured parent lessons, setting reading goals, and 6 children's books (one mailed home each week), and options to receive weekly reminders (e.g., email or text) to encourage reading readiness.
  Arms: weLearn2Read

SUMMARY:
This study will include 12 rural Head Start programs, randomly assigned to one of two groups: weSIPsmarter vs. control. The main goal is to find out if weSIPsmarter helps reduce sugary drink consumption in preschool-aged children and their parents.

DETAILED DESCRIPTION:
Sugary drinks are the largest single source of calories in the US diet and contribute approximately 8% and 7% of total energy intake for US youth and adults, respectively. Unfortunately, the prevalence of daily sugary drink intake is significantly higher in nonmetropolitan US counties, relative to metropolitan counties (adjusted prevalence ratio = 1.32). Also, an estimated 47% of children age 2-5 consume sugary drinks daily. High sugary drink intake contributes to the development of numerous chronic conditions, including cancer. Despite convincing data on risky sugary drink behaviors in rural counties and among preschool-aged children, there are substantial gaps in the intervention literature. For example, few sugary drink interventions have targeted the needs of US rural regions, few have effectively used scalable technology to reduce child's sugary drinks, and most fail to report on external validity factors. This research addresses these needs and builds on the research team's extensive digital Health expertise and successful sugary drink research within rural communities. Head Starts across defined rural areas (i.e., RUCC 4-9) in Appalachia and the southern Black Belt will be included. The intervention targets parents as the agent of change and aims to improve parent-child dyad outcomes. Phase 1 is guided by the Adaptome framework. In partnership with rural Head Start staff and parents, a user-centered design process will be applied to adapt an existing evidence-based sugary drink interventions to a digital intervention. This new program, called weSIPsmarter, will be a highly interactive, structured program consisting of multiple evidence-based behavioral change components, including use of ecological momentary assessment (EMA) to encourage self-monitoring of beverage behaviors and parenting feeding practices, action planning, a resource help line, and drinking water vouchers for families with concerns related to in-home tap water quality. Phase 2 is guided by RE-AIM and includes a 2 group cluster RCT design [weSIPsmarter vs. control] with 3 assessment (pre, 9-week post, and 12-month follow-up) periods. Twelve Head Start center clusters with an average of 31 parent-child dyads per cluster (total of 372 parent-child dyads) will be randomized. It is hypothesized that weSIPsmarter will be more efficacious at reducing sugary drink consumption than control. Changes in secondary outcomes will also be evaluated, including parent-child dyad outcomes (e.g., diet quality, water, BMI, QOL, behavioral theory constructs) and maintenance at 12-months post intervention. Additional secondary aims will examine reach, describe parent engagement, and apply a mixed-methods process evaluation to evaluate adoption and implementation among Head Starts. Mediators and moderators (e.g., social determinant of health indicators) to engagement and efficacy outcomes will be explored, along with organizational-level maintenance. The long-term goal of this primary prevention research is to develop an efficacious sugary drink reduction intervention that has high reach among rural, low socioeconomic, children ages 2-5 and their parents.

ELIGIBILITY:
Inclusion Criteria:

1. Head Start sites: Head Start sites will be located in or adjacent to a rural county (RUCC 4-9), fall within the planned Appalachia and Black Belt regions, have an enrollment of 120 families or more, and exhibit commitment and capacity to the scope of work.
2. Participants: Children enrolled must be between the ages of 2 and 5 year, be enrolled in a participating Head Start, and have a legal guardian ("parent," able under law to consent for their child to participate) who has enrolled in the trial themselves and provided consent for the child. Only one parent-child dyad per household is eligible to participate in the trial.

Exclusion Criteria:

* Parents could not have participated in formative work for this study completed under SBS 4522.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 744 (Estimated)
Dates: Start 2025-08-06 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Child sugar-sweetened beverage (SSB) ounces | Baseline and 9 weeks
  The Beverage Intake Questionnaire for Preschool-aged Children (BEVQ-PS) assesses the intake of sugar-sweetened beverages (SSBs) by measuring the frequency and amount (in ounces) across beverage categories. The ounces are then then aggregated to calculate the total SSB intake in ounces.

SECONDARY OUTCOMES:
Child sugar sweetened beverage (SSB) ounces | 12 month
  The Beverage Intake Questionnaire for Preschool-aged Children (BEVQ-PS) assesses the intake of sugar-sweetened beverages (SSBs) by measuring the frequency and amount (in ounces) across beverage categories. The ounces are then then aggregated to calculate the total SSB intake in ounces.
Parent sugar-sweetened beverage (SSB) ounces | Baseline, 9 weeks, 12 months
  The Beverage Intake Questionnaire (BEVQ-15) assesses the intake of sugar-sweetened beverages (SSBs) by measuring the frequency and amount (in ounces) across beverage categories. The ounces are then then aggregated to calculate the total SSB intake in ounces.
Child Weight in pounds | Baseline, 9 weeks, 12 months
  Measured using a cellular enabled in-home BodyTrace digital scale
Child Height in feet and inches | Baseline, 9 weeks, 12 months
  Measured via stadiometer
Child Body Mass Index (BMI) Percentile | Baseline, 9 weeks, 12 months
  Child's Body Mass Index (BMI) will be calculated using the standard formula: weight(kg)/height(m)2. BMI z-score will be calculated using CDC growth charts and converted to BMI-for-age percentile based on CDC growth charts for children and teens ages 2 through 19.
Parent Weight in pounds | Baseline, 9 weeks, 12 months
  Measured using a cellular enabled in-home BodyTrace digital scale.
Parent Height in feet and inches | Baseline
  Self-reported
Parent Body Mass Index (BMI) | Baseline, 9 weeks, 12 months
  Parent's Body Mass Index (BMI) will be calculated using the standard formula: weight(kg)/height(m)2.
Parent number of unhealthy days | Baseline, 9 weeks, 12 months
  The number of unhealth days, a measure of Quality of Life (QOL), will be assessed using Center's for Disease Control Healthy Day module. Higher number of days means worse outcome.
Proportion of parents with limited health literacy | Baseline, 9 weeks, 12 months
  Assessed using the Newest Vital Sign. Scores range from 0-6 with 0-4 considered limited health literacy and 5-6 considered to be adequate health literacy.
Parent sugary-sweetened beverage (SSB) media literacy score | Baseline, 9 weeks, 12 months
  Measured with sugary-sweetened beverage (SSB) media literacy instrument which includes 6 items measured on a 7-point Likert scale (1, strongly disagree; 7, strongly agree). Scores range from 7-42; Higher scores equate to higher SSB media literacy.
eHealth digital literacy score | Baseline, 9 weeks, 12 months
  The eHEALS digital literacy test is an 8-item measure of eHealth literacy developed to measure the participants combined knowledge, comfort and perceived skills at finding, evaluating and applying electronic health information to health problems. The test is measured with a 5-point Likert scale with response options ranging from "strongly disagree" to "strongly agree." Total scores of the eHEALS are summed to range from 8 to 40, with higher scores representing higher self-perceived eHealth literacy.
Division of Responsibility (DOR) feeding approach score | Baseline, 9 weeks, 12 months
  Assessed using Satter Parent-Child Feeding Measure (sDOR.2-6y™). Includes 12 times, with scores ranging from 0-32. Higher scores indicate greater adherence to the Division of Responsibility (DOR) feeding approach.
Frequency of sugar-sweetened beverages (SSB) in the home | Baseline, 9 weeks, 12 months
  Home availability of 7 categories of sugar sweetened beverages (SSB) in the home. Responses are on a 5-point Likert scale (1, never; 5, always). Scores range from 7-35, with higher scores meaning higher home availability of SSB.
Child fruits and vegetables (cup equivalents per day) | Baseline, 9 weeks, 12 months
  Assessed using the Dietary Screener Questionnaire (DSQ). Validated scoring algorithms are used to convert frequency of food items into fruits and vegetables cup equivalents per day.
Child added sugars (teaspoon equivalents per day) | Baseline, 9 weeks, 12 months
  Assessed using the Dietary Screener Questionnaire (DSQ). Validated scoring algorithms are used to convert frequency of food items into added sugars teaspoon equivalents per day.
Child added sugars from sugar-sweetened beverages (teaspoon equivalents per day) | Baseline, 9 weeks, 12 months
  Assessed using the Dietary Screener Questionnaire (DSQ). Validated scoring algorithms are used to convert frequency of food items into added sugars from sugar-sweetened beverages teaspoon equivalents per day.
Child dairy (cup equivalents per day) | Baseline, 9 weeks, 12 months
  Assessed using the Dietary Screener Questionnaire (DSQ). Validated scoring algorithms are used to convert frequency of food items into dairy cup equivalents per day.
Child whole grains (ounce equivalents per day) | Baseline, 9 weeks, 12 months
  Assessed using the Dietary Screener Questionnaire (DSQ). Validated scoring algorithms are used to convert frequency of food items into whole grains ounce equivalents per day.
Child calcium (milligrams per day) | Baseline, 9 weeks, 12 months
  Assessed using the Dietary Screener Questionnaire (DSQ). Validated scoring algorithms are used to convert frequency of food items into calcium milligrams per day.
Child fiber (grams per day) | Baseline, 9 weeks, 12 months
  Assessed using the Dietary Screener Questionnaire (DSQ). Validated scoring algorithms are used to convert frequency of food items into fiber grams per day.
Child red meat (times per day) | Baseline, 9 weeks, 12 months
  Assessed using the Dietary Screener Questionnaire (DSQ). Validated scoring algorithms are used to convert frequency of food items into red meat times per day.
Child processed meat (times per day) | Baseline, 9 weeks, 12 months
  Assessed using the Dietary Screener Questionnaire (DSQ). Validated scoring algorithms are used to convert frequency of food items into processed meat times per day.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Christiansburg, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
All the deidentified behavioral-related data (as described it the outcome measure section) will be achieved in the University of Virginia's data repository, LibraData. The clinical trial outcome data will be findable and identifiable in LibraData via a persistent identifier (DOI), which is created for each LibraData dataset.